# **RTOG FOUNDATION**

# **RTOG 3502**

(ClinicalTrials.gov NCT #: 01753414)

POSTILV: A RANDOMIZED PHASE II TRIAL IN <u>P</u>ATIENTS WITH <u>O</u>PERABLE <u>ST</u>AGE <u>I</u> NON-SMALL CELL <u>L</u>UNG CANCER: RADICAL RESECTION <u>V</u>ERSUS ABLATIVE STEREOTACTIC RADIOTHERAPY

Amendment 2: August 6, 2018

# **Informed Consent (English Language)**

Sponsor / Study Title: RTOG Foundation of American College of Radiology/

"POSTILV: A Randomized Phase II Trial in Patients with Operable Stage I Non-Small Cell Lung Cancer: Radical Resection Versus Ablative Stereotactic

Radiotherapy"

Protocol Number: RTOG 3502

**Principal Investigator:** 

(Study Doctor)

«PiFullName»

Telephone: «IcfPhoneNumber»

Address: «PiLocations»

This is a clinical trial, a type of research study. Your study doctor will explain the clinical trial to you. Clinical trials include only people who choose to take part. Please take your time to make your decision about taking part. You may discuss your decision with your friends and family. You can also discuss it with your health care team. If you have any questions, you can ask your study doctor for more explanation.

You are being asked to take part in this study because you have lung cancer that may be removed by surgery.

### Why is this study being done?

The standard treatment for your type of cancer is surgery.

The purpose of this study is to compare surgery to stereotactic body radiation therapy (SBRT) to see the effects these treatments have on you and your lung cancer. SBRT may have fewer side effects than surgery, but we do not know if SBRT is as effective at removing your cancer or preventing it from returning.

SBRT is a newer radiation treatment that gives fewer but higher and possibly more effective doses of radiation than standard radiation. The technique of giving a higher effective dose per treatment may work better to kill cancer cells potentially with fewer side effects than standard radiation therapy. SBRT uses special equipment to position the patient and guide focused x-ray beams toward the cancer and away from normal lung tissue. Research so far suggests that SBRT can reduce the size or eventually eliminate lung tumors effectively and is relatively safe for lungs and other organs in your body.

### How many people will take part in the study?

About 76 people will take part in this study.

# What will happen if I take part in this research study?

You will have a PET/CT scan to see if you can take part in this study. If the scan shows that you cannot take part, your doctor will talk with you about other treatments.

If the scan shows that you can take part in the study, you will be "randomized" into one of the study groups described below. Randomization means that you are put into a group by chance. A computer program will place you in one of the study groups. Neither you nor your study doctor can choose the group you will be in. You will have an equal chance of being placed in one of the groups.

If you are in group 1 (often called "Arm A"): You will have surgery to remove all or most of the lung cancer and one lobe (section) of the lung.

If you are in group 2 (often called "Arm B"): You will have SBRT, once every other day for 5 treatments.

<u>Before SBRT begins</u>, you will have a treatment planning session. You will lie in a specific position, possibly within a frame device or on a large plastic bag filled with tiny foam balls similar to a bean bag. The purpose of the frame or bag is to hold your body as still as possible for planning and treatment. After you are positioned, doctors will check your breathing and see how your tumor and organs move. The doctors will try to limit the effect of that movement on the position of your tumor by timing your breathing. They may use a device to control the depth of your breathing or one to monitor the rate and pattern of your breathing so that they will be able to deliver the radiation to the tumor while accounting for the effect of breathing.

Radiation Treatment: Usually 7-10 days after the radiation planning session, you will return to the radiation medicine department for your radiation treatment. For your treatment, you will lie in the device that was used for your planning session. You will lie as still as possible and breathe normally (or have your breathing controlled by a device) while your radiation is delivered. It will take approximately one to two hours to deliver the radiation. During the process of radiation, participants can become claustrophobic. Medications can be given to make you feel more comfortable should this happen. Also, your doctor may give you pain medication before each treatment to decrease any discomfort you may have due to laying on a hard surface and/or due to laying with your arms held above your head during the treatment.

### Before you begin the study:

You will need to have the following exams, tests or procedures to find out if you can be in the study. These exams, tests or procedures are part of regular cancer care and may be done even if you do not join the study. If you have had some of them recently, they may not need to be repeated. This will be up to your study doctor.

- Physical examinations by several doctors
- Checking your weight
- Evaluation of your ability to carry out daily activities
- A PET (Positron Emission Tomography) scan of your body: A small amount of radioactive material is injected into your vein, and a scanner makes a detailed picture of areas inside your body
- A CT (Computed Tomography) scan of your lungs and abdomen with contrast: a CT scan is a study using x-rays to look at one part of your body. Contrast means that dye is injected into your vein to increase the differences between normal and abnormal tissue.
- Tests of your breathing and lung function
- For women who are able to have children, a test to see that they are not pregnant
- Endobronchial Ultrasound: A tube is inserted through your mouth or nose in the
  airway leading to your lungs. After the tube is in place, the doctor uses a probe to
  send sound waves into the lungs to make an image. To obtain tissue or fluids
  from the lungs, the doctor uses a small needle or probe. This procedure may
  require you to have anesthesia.

# **During the study:**

If the exams, tests and procedures show that you can be in the study, and you choose to take part, then you will need the following tests and procedures. They are part of regular cancer care.

<u>For Group 2 patients after SBRT is completed</u>: Evaluation of any side effects from treatment you may be having

## 4-6 weeks after surgery or SBRT

- Physical examinations by several doctors
- Checking your weight
- Evaluation of your ability to carry out daily activities
- Evaluation of any side effects from treatment you may be having

### For Group 1 patients, 4-6 weeks after surgery

- A CT (Computed Tomography) scan of your lungs and abdomen with contrast
- A PET (Positron Emission Tomography) scan of your body

### You will need these tests and procedures in follow-up visits:

At 3, 6, 9, 12, 18, 24 and 36 months after treatment: A CT (Computed Tomography) scan of your lungs and abdomen with contrast

At 3, 12, and 24 months after treatment: A PET (Positron Emission Tomography) scan of your body

Every 3 months for years 1-2 years, every 6 months for year 3, then yearly for your lifetime:

- Physical examination
- Checking your weight
- Evaluation of your ability to carry out daily activities
- Evaluation of any side effects from treatment you may be having
- If your doctor recommends, tests of your breathing and lung function

## **Study Plan**

Another way to find out what will happen to you during the study is to read the chart below. Start reading at the top and read down the list, following the lines and arrows.



### How long will I be in the study?

Group 1 patients will receive surgery. Group 2 patients will receive 1 SBRT treatment every other day for 5 treatments.

After your treatment is completed, you will be seen in follow-up visits every 3 months for years 1-2 years, every 6 months for year 3, then once a year for 2 years, for a total of 5 years of follow up from the time you begin treatment.

### Can I stop being in the study?

Yes. You can decide to stop at any time. Tell the study doctor if you are thinking about stopping or decide to stop. He or she will tell you how to stop safely.

It is important to tell the study doctor if you are thinking about stopping so any risks from the surgery or SBRT can be evaluated by him/her. Another reason to tell your study doctor that you are thinking about stopping is to discuss what follow-up care and testing could be most helpful for you.

The study doctor may stop you from taking part in this study at any time if he/she believes it is in your best interest; if you do not follow the study rules; or if the study is stopped.

## What side effects or risks can I expect from being in the study?

You may have side effects while on the study. Everyone taking part in the study will be watched carefully for any side effects. However, researchers don't know all the side effects that may happen. Side effects may be mild or very serious. Your health care team may give you medicines to help lessen side effects. Many side effects go away soon after surgery or SBRT. In some cases, side effects can be serious, long lasting, or may never go away. There also is a risk of death.

You should talk to your study doctor about any side effects that you have while taking part in the study.

# Risks and side effects related to lung surgery

### <u>Likely</u>

- Prolonged chest tube drainage after surgery
- Persistent cough or trouble breathing that may require further treatment
- Shortness of breath

### Less Likely

- Lung infection/pneumonia
- A blood clot in the lung
- A blood clot in a large vein, which could result in a stroke or a heart attack in some cases
- Prolonged need for a tube placed in your airway to help you breath during the surgery for longer than 24 hours after surgery is finished or
- Replacing the tube in your airway after it is initially taken out
- Wound infection
- Leakage of air from the lung after your lung cancer has been removed
- Injury to the nerves of your voice box (larynx), which may result in hoarseness or difficulty swallowing
- Changes in tests that show how your lungs are working

### **Rare but Serious**

- Sepsis (a severe form of infection)
- Heart attack
- Irregular or rapid heartbeat
- Severe inflammation of the lung, which can affect your ability to breath normally
- Injury to a blood vessel that can result in heavy bleeding during or after surgery

#### Risks and side effects related to the SBRT

### Likely

- Damage to surrounding normal lung and/or collapse of a portion of treated lung
- Changes in the lungs as the tumor shrinks; these changes will be recognized by your radiation doctor on your x-rays or scans as expected "scarring" that is developing. In most patients, no noticeable symptoms will result from this lung damage.
- Fatigue
- Redness of irritation of the skin in the treatment
- Hair loss in the treatment area (chest hair)
- Some soreness of the ribs with an increased risk of rib fracture. Treatment for such symptoms usually consists of rest, heat, and pain medication.

### Less Likely

- Cough
- Increased phlegm production
- Difficulty breathing
- Fever

#### Rare but Serious.

- Some patients can have the following symptoms associated with lung scarring: shortness of breath, cough, fever, and/or pain in the chest wall. These patients may require oxygen for a short time or permanently. Lung damage can be life threatening.
- Damage to the lining of the heart, which can cause fluid accumulation around the heart and chest pain, shortness of breath, and/or irregular or rapid heart beat
- Damage to the heart muscle, which can cause heart attack, heart failure, or death
- Damage to the spinal cord, which can cause numbness, weakness, tingling, and/or inability to use the arms and/or legs
- Damage to the esophagus, which can cause problems with swallowing
- Damage to the large blood vessels surrounding the heart, which could cause coughing up of blood and possibly death
- Severe pain or skin damage leading to an open wound

During the process of treatment planning and radiation, you will lie in a specific position, possibly within a frame device, and some patients can become claustrophobic. Medications can be given to make you feel more comfortable should this happen. Also, your doctor may give you pain medication before each treatment to decrease any discomfort you may have due

to laying on a hard surface and/or due to laying with your arms held above your head during the treatment.

### Reproductive risks:

This study may be harmful to a nursing infant or an unborn child. If you are a woman able to have children and have not been surgically sterilized (tubal ligation or hysterectomy), you must have a pregnancy test before enrolling in this study. If you are unwilling to use adequate birth control measures to prevent pregnancy, you should not participate in this study. If you should become pregnant while you are on this study, you must tell your doctor immediately.

If you are a man able to father children, the treatment you may receive may risk harm to an unborn child unless you use a form of birth control approved by your doctor. If you are unwilling to use adequate birth control measure to prevent pregnancy you should not participate in this study. If you suspect you have caused anyone to become pregnant while you are on this study, you must tell your doctor immediately.

For more information about risks and side effects, ask your study doctor.

# Are there benefits to taking part in the study?

Taking part in this study may or may not make your health better. While researchers hope the study will help determine if SBRT is as effective as surgery in treating lung cancer, with less side effects. We do know that the information from this study will help researchers learn more about SBRT as a treatment for cancer. This information could help future cancer patients.

# What other choices do I have if I do not take part in this study?

Your other choices may include:

- Getting treatment or care for your cancer without being in a study
- Taking part in another study
- Getting no treatment

Talk to your study doctor about your choices before you decide if you will take part in this study.

## Will my medical information be kept private?

Data are housed at RTOG Headquarters in a password-protected database. We will do our best to make sure that the personal information in your medical record will be kept private. However, we cannot guarantee total privacy. Your personal information may be given out if required by law. If information from this study is published or presented at scientific meetings, your name and other personal information will not be used.

Organizations that may look at and/or copy your medical records for research, quality assurance, and data analysis include:

- The Radiation Therapy Oncology Group (RTOG)
- China POSTILV Trial Group
- The Institutional Review Boards (IRB) associated with this study. The IRBs are groups
  of people who review the research with the goal of protecting the people who take part
  in the study.

# What are the costs of taking part in this study?

[Participating institutions: Insert your standard language here regarding health coverage for your patients (e.g. National health plan).]

You will not be paid for taking part in this study.

| What happens if I am inj | ured because I took | part in this study | <b>y?</b> |
|---|---|---|---|
|---|---|---|---|

| It is important that you tell your study doctor,<br>you feel that you have been injured because of taki<br>doctor in person or call him/her at | [investigator's name(s)], if ng part in this study. You can tell the study [telephone number]. |
|---|---|
| You will get medical treatment if you are injured as and/or your health plan will be charged for this trea | 0 1 |

# What are my rights if I take part in this study?

Taking part in this study is your choice. You may choose either to take part or not to take part in the study. If you decide to take part in this study, you may leave the study at any time. No matter what decision you make, there will be no penalty to you and you will not lose any of your regular benefits. Leaving the study will not affect your medical care. You can still get your medical care from our institution.

We will tell you about new information or changes in the study that may affect your health or your willingness to continue in the study.

A Data Monitoring Committee (DMC) will be regularly meeting to monitor safety and other data related to this study. The Committee members may receive confidential patient information, but they will not receive your name or other information that would allow them to identify you by name.

In the case of injury resulting from this study, you do not lose any of your legal rights to seek payment by signing this form.

treatment.

# Who can answer my questions about the study?

| You can talk to your study doctor about any qu | uestions or concerns you have about this study. |
|---|---|
| Contact your study doctor | [name(s)] at |
| [telephone number]. | |
| For questions about your rights while taking pa | art in this study, call the |
| [name of cente | r] Institutional Review Board (a group of people |
| who review the research to protect your rights | ) at (telephone number). |
| [Note to Local Investigator: Contact informatio | n for patient representatives or other individuals |
| in a local institution who are not on the IRB or | research team but take calls regarding clinical |
| trial questions can be listed here.] | |

Please note: This section of the informed consent form is about additional research that is being done with people who are taking part in the main study. You may take part in this additional research if you want to. You can still be a part of the main study even if you say 'no' to taking part in this additional research.

You can say "yes" or "no" to each of the following studies. Below, please mark your choice for each study.

### Consent Form for Use of Tissue and Blood for Research

<u>[Institutions participating in the trial</u>: The text below is sample text only. Add site-specific language for specimen collection as necessary.]

### **About Using Tissue and Blood for Research**

You are going to have or have had a biopsy to see if you have cancer. Your doctor will remove some body tissue to do some tests. The results of these tests will be given to you by your doctor and will be used to plan your care.

We would like to keep some of the tissue that is left over for future research.

In addition to the tumor tissue, we would like to collect 3-4 teaspoons of your blood at the following time points: For Group 1 patients before surgery, during surgery, before you leave the hospital, and 4-6 weeks after surgery; for Group 2 patients before the first radiation treatment, after the third radiation treatment, immediately after treatment, and 4-6 weeks after treatment.

If you agree, this tissue and blood will be kept and may be used in research to learn more about cancer and other diseases.

Your tissue and blood may be helpful for research whether you do or do not have cancer. The research that may be done with your tissue and blood is not designed specifically to help you. It might help people who have cancer and other diseases in the future.

Reports about research done with your tissue and blood will not be given to you or your doctor. These reports will not be put in your health record. The research will not have an effect on your care.

# **Things to Think About**

The choice to let us keep the left over tissue and blood for future research is up to you. No matter what you decide to do, it will not affect your care or your participation in the main part of the study.

If you decide now that your tissue and blood can be kept for research, you can change your mind at any time. Just contact us and let us know that you do not want us to use your tissue and blood. Then any tissue and blood that remains will no longer be used for research and will be returned to the institution that submitted it.

In the future, people who do research may need to know more about your health. While the doctor/institution may give them reports about your health, it will not give them your name, address, phone number, or any other information that will let the researchers know who you are.

Sometimes tissue and blood is used for genetic research (about diseases that are passed on in families). Even if your tissue and blood is used for this kind of research, the results will not be put in your health records.

Your tissue and blood will be used only for research and will not be sold. The research done with your tissue and blood may help to develop new treatments for cancer in the future.

#### **Benefits**

The benefits of research using tissue and blood include learning more about what causes cancer and other diseases, how to prevent them, and how to treat them.

#### **Risks**

The greatest risk to you is the release of information from your health records. We will do our best to make sure that your personal information will be kept private. The chance that this information will be given to someone else is small.

# **Making Your Choice**

| Please read each sentence below and think about your choice. After reading each sentence, circle "Yes" or "No". If you have any questions, please talk to your doctor or nurse, or call our research review board at [IRB's phone number]. |
|---|
| No matter what you decide to do, it will not affect your care. |
| <ul> <li>1. My specimens may be kept for use in research to learn about, prevent, or treat cancer, as follows:</li> <li>Tissue □Yes □ No</li> <li>Blood □Yes □ No</li> </ul> |
| <ul> <li>2. My specimens may be kept for use in research to learn about, prevent or treat other health problems (for example: diabetes, Alzheimer's disease, or heart disease), as follows:</li> <li>Tissue □Yes □ No</li> <li>Blood □Yes □ No</li> </ul> |
| <ol> <li>Someone may contact me in the future to ask me to take part in more research.</li> <li>□Yes</li> <li>□ No</li> </ol> |
| You will get a copy of this form. If you want more information about this study, ask your study doctor. |
| Signature |
| I have been given a copy of all [insert total of number of pages] pages of this form. I have read it or it has been read to me. I understand the information and have had my questions answered. I agree to take part in this study. |
| Participant |
| Date |